CLINICAL TRIAL: NCT01509534
Title: Guideline-based Pacing Therapy for Reflex Syncope
Acronym: SUP2
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Multidisciplinare per lo Studio della Sincope (Other)
Responsible Party: Sponsor
Other Study IDs: GIMSI-001-2011
Record Dates: First submitted 2011-12-05; First posted 2012-01-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Syncope
Keywords: pacemaker; implantable loop recorder; syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study hypothesis: Dual-chamber pacemaker therapy with rate-hysteresis features is effective in preventing syncopal recurrences in patients affected by cardioinhibitory (CI) forms of reflex syncope diagnosed by means of carotid sinus massage, tilt table testing or implantable loop recorder (ILR). The outcome is measured either by the time to first syncopal recurrence or the total syncope burden.

DETAILED DESCRIPTION:
Background Divergence of opinion exists regarding the efficacy of cardiac pacing in patients affected by different forms of reflex syncope.

Definitions.

Severe syncope is defined when:

* it is perceived by patient that it alters his/her quality of life, and
* is unpredictable because occurs without, or with very short prodromes < 10 sec (thus exposing patients to risk of trauma) or, if preceded by prodromes, syncope recurs despite appropriate therapies (CPM or drugs).

Recurrent syncopes: at least 2 episodes during the last year (including the index episode) or 3 episodes during the last 2 years (including the index episode).

Suspected (undetermined) reflex syncope: the suspicion of reflex syncope is based on a history of uncertain syncope in the absence of (i) severe structural heart disease, significant ECG abnormalities, or rhythm disturbances; (ii) orthostatic hypotension; and (iii) non-syncopal causes of transient loss of consciousness.

Study protocol

1. The eligible patients undergo firstly carotid sinus massage (according to the method of symptoms); if a diagnosis of cardioinhibitory carotid sinus syndrome (CI-CSS) is made, a pacemaker is implanted and follow-up immediately starts.
2. If the carotid sinus massage is negative or vasodepressor, the patients undergo tilt table testing (with nitroglycerin or clomipramine drug challenge); if a diagnosis of VASIS 2B form is made, a pacemaker is implanted and follow-up immediately starts.
3. If tilt table testing is negative or a form different from VASIS 2B is induced, the patients undergo ILR implantation. If a diagnosis of asystolic reflex syncope is made, a pacemaker is implanted and follow-up immediately starts.

End-points End-point of the study is syncope recurrence after pacemaker (PM) implantation. Syncope is defined as complete transient loss of consciousness. Pre-syncope is counted but it is not an end-point.

Primary end-points:

1. Comparison of the time to first syncopal recurrence in CI-CSS and CI-TTT pts with PM and in control patients with ILR.
2. Intra-patient comparison of the syncope burden in the year before and in the year following PM implant in all patients receiving a PM (CCS, TTT and ILR groups). Index syncope is not counted.

Follow-up One year after PM implantation for all enrolled patients for burden of syncope end-points Until the study end for time to first syncope recurrence end-points. Thus, the study ends one year after the enrollment of the last patient.

Study size Based on the sample size calculation the study will stop when 700 patients are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by severe, recurrent, certain or suspected (undetermined) reflex syncopes, aged ≥ 40 years.

Exclusion Criteria:

* Reflex syncopes due to reversible causes, e.g., vasoactive drugs, concomitant diseases, etc
* Suspected of certain cardiac syncope
* Syncope caused by orthostatic hypotension
* Non-syncopal causes of transient loss of consciousness

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by reflex syncopes
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
syncope recurrence after PM implantation | 1 year

SECONDARY OUTCOMES:
syncope burden after PM implantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Ospedali del Tigullio, Lavagna, Italy
Locations (8):
- Italy (8):
  - Ospedale Generale Regionale, Bolzano
  - AO di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - PO S. Giuseppe, Empoli
  - AO Careggi, Florence
  - Nuovo Ospedale S. Giovanni di Dio, Florence
  - Department of Cardiology, Ospedali del Tigullio, Lavagna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale SS. Annunziata, Taranto

REFERENCES:
- [Derived] Solari D, Tesi F, Unterhuber M, Gaggioli G, Ungar A, Tomaino M, Brignole M. Stop vasodepressor drugs in reflex syncope: a randomised controlled trial. Heart. 2017 Mar;103(6):449-455. doi: 10.1136/heartjnl-2016-309865. Epub 2016 Sep 23. PMID 27664002
- [Derived] Brignole M, Arabia F, Ammirati F, Tomaino M, Quartieri F, Rafanelli M, Del Rosso A, Rita Vecchi M, Russo V, Gaggioli G; Syncope Unit Project 2 (SUP 2) investigators. Standardized algorithm for cardiac pacing in older patients affected by severe unpredictable reflex syncope: 3-year insights from the Syncope Unit Project 2 (SUP 2) study. Europace. 2016 Sep;18(9):1427-33. doi: 10.1093/europace/euv343. Epub 2015 Nov 26. PMID 26612880
- [Derived] Brignole M, Ammirati F, Arabia F, Quartieri F, Tomaino M, Ungar A, Lunati M, Russo V, Del Rosso A, Gaggioli G; Syncope Unit Project (SUP) Two Investigators. Assessment of a standardized algorithm for cardiac pacing in older patients affected by severe unpredictable reflex syncopes. Eur Heart J. 2015 Jun 21;36(24):1529-35. doi: 10.1093/eurheartj/ehv069. Epub 2015 Mar 29. PMID 25825044